CLINICAL TRIAL: NCT02341274
Title: Effects of Altered Formulation on the Bioequivalence of Tacrolimus in Healthy Female and Male Volunteers
Brief Title: Effects of Altered Formulation on the Bioequivalence of Tacrolimus in Healthy Female and Male Volunteeers
Acronym: ASDBioequiv
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1409250017
Record Dates: First submitted 2015-01-07; First posted 2015-01-19 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2017-09

CONDITIONS: Bioequivalence
Keywords: Tacrolimus; Drug Formulation; Absorption; Bioavailability; Healthy Volunteer
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fresh Brand Name Tacrolimus (Prograf®) (Active Comparator): Oral administration of 5 mg capsule of fresh brand name tacrolimus (Prograf®) to healthy volunteer on an empty stomach. Blood samples will be collected from the indwelling venous catheter (∼10 ml) after 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours after dosing. The volunteers will be allowed to eat a normal lunch 3 hours after taking their tacrolimus dose. After the 24-hour blood sample has been collected, the volunteer will be discharged.
  Interventions: Drug: Tacrolimus
- Fresh Generic Tacrolimus (Active Comparator): Oral administration of 5 mg capsule of fresh generic tacrolimus to healthy volunteer on an empty stomach. Blood samples will be collected from the indwelling venous catheter (∼10 ml) after 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours after dosing. The volunteers will be allowed to eat a normal lunch 3 hours after taking their tacrolimus dose. After the 24-hour blood sample has been collected, the volunteer will be discharged.
  Interventions: Drug: Tacrolimus
- Low Crystal Generic Tacrolimus (Active Comparator): Oral administration of 5 mg capsule of 10-30% crystallized generic tacrolimus (Low Crystal) to healthy volunteer on an empty stomach. Blood samples will be collected from the indwelling venous catheter (∼10 ml) after 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours after dosing. The volunteers will be allowed to eat a normal lunch 3 hours after taking their tacrolimus dose. After the 24-hour blood sample has been collected, the volunteer will be discharged.
  Interventions: Drug: Tacrolimus
- High Crystal Generic Tacrolimus (Active Comparator): Oral administration of 5 mg capsule of 40-60% crystallized generic tacrolimus (High Crystal) to healthy volunteer on an empty stomach. Blood samples will be collected from the indwelling venous catheter (∼10 ml) after 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours after dosing. The volunteers will be allowed to eat a normal lunch 3 hours after taking their tacrolimus dose. After the 24-hour blood sample has been collected, the volunteer will be discharged.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Bioequivalence study
  Other Names: FK-506, FK506, D016559, WM0HAQ4WNM

SUMMARY:
Amorphous solid dispersion (ASD) formulations are increasingly used by the pharmaceutical industry to develop poorly water-soluble drugs into effective oral dosage forms. Examples include the antifungal drug itraconazole, the HIV protease inhibitor combination, lopinavir/ritonavir and the immunosuppressive, tacrolimus. There is potential for significant variation in bioavailability of ASD and thus heightened concern regarding the therapeutic efficacy as generic versions of these poorly water-soluble compounds become approved. The variation in bioavailability is to be expected because of our limited understanding of the precise physical chemistry of drug polymer amorphous solid dispersion formulations.

DETAILED DESCRIPTION:
The specific aim is to conduct a randomized, single dose, four-treatment, four-period cross-over bioequivalence (BE) study in 24 healthy normal adult volunteers (males and non-gravid females) to evaluate the in vivo performance of fresh and aged brand name and generic amorphous solid dispersion (ASD) preparations of tacrolimus. The pharmacokinetics of tacrolimus as fresh Prograf® and aged Prograf®, fresh generic tacrolimus capsules and aged generic tacrolimus capsule will be determined and compared in healthy volunteers. The hypothesis to be tested is that the tacrolimus in the amorphous solid dispersion formulation will be partially crystalized upon treatment with controlled heat and humidity and will demonstrate lower absorption (lower relative bioavailability) compared to the fresh product. Moreover, the expectation is that the heat- and humidity-stressed generic formulations will not be robust to crystallization as the stressed brand name drug and will demonstrate a decreased in vivo performance and loss of bioequivalence.

A total of 24 healthy female and male volunteers (age 18 to 49 years old) will be recruited to participate in this study. Volunteers will be determined to be free of significant medical conditions as assessed by medical history, physical examination, and blood and urine tests. Volunteers will be randomly allocated to receive one of the four treatment sequence groups and, on each occasion, receive one of the following: Fresh Prograf (RLD), fresh generic tacrolimus, 10-30% crystallized generic (Low Crystal), and 40-60% crystallized generic (High Crystal) tacrolimus. There will be a minimum 2-week washout between treatments. On each occasion, healthy volunteers will be administered tacrolimus, 5 mg, as a single capsule orally on an empty stomach with approximately 240 mL of water. Blood samples will be collected from the indwelling venous catheter (∼10 ml) after 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours after dosing. Subjects will be regularly monitored during this time. The volunteers will be allowed to eat a normal lunch 3 hours after taking their tacrolimus dose.

The primary endpoints will be the maximum blood concentration (Cmax) and the area under the curve (AUC) from zero to 24 hours and the AUC extrapolated from zero to infinity for tacrolimus for this bioequivalence study as recommended by the FDA guidance for industry. We will compute the AUC (from zero to 24 hours) to the last time point with measurable concentration using the linear trapezoidal rule and the AUC from time zero to time infinity with extrapolation computed as the quotient of the last measurable concentration and the terminal slope of the log concentration vs. time curve. In addition, we will report half-life of tacrolimus estimated from the terminal slope of the concentration vs. time plot determined by linear least squares regression. The peak blood tacrolimus concentration (Cmax,) and the time to Cmax (Tmax,) will be determined by visual inspection of the individual subject concentration-time curves.

A treatment will be considered bioequivalent if the geometric least square mean ratios and 90% confidence interval for Cmax and AUC fall between 0.80 to 1.25 of the fresh Prograf®.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 49 years old.
* Healthy individuals without any significant medical condition.
* Nonsmoker or individuals willing to refrain from smoking or use of tobacco or marijuana for at lest one month prior to and until the completion of the study. The entire study for each volunteer will last for minimum of 42 days.
* Ability to commit the time requested for this study.
* Ability to swallow capsules.

Exclusion Criteria:

* Underweight (weigh less than 52 kg or 114 lb.) or overweight (body mass index (BMI) greater than 32).
* History or current alcohol or drug abuse (more than 3 alcoholic drinks per day on a regular basis).
* History or current significant health conditions such as heart, liver, or kidney.
* History or current psychiatric illness such as depression, anxiety, or nervousness.
* History or current gastrointestinal disorders such as persistent diarrhea or malabsorption that would interfere with the absorption of orally administered drugs.
* Individuals having a serious infection within the last month.
* Donation of blood within the past two months.
* Blood hemoglobin less than 12.5 mg/dL.
* Individuals who are regularly taking prescriptions, over-the-counter, herbal or dietary supplements, alternative medications, or hormonal agents (i.e. oral contraceptives, intra-uterine device with hormones).
* Females with a positive pregnancy test.
* Breastfeeding.
* Females of child-bearing potential who are unable or unwilling to either practice abstinence or to use two non-hormonal forms of birth control (e.g. condom, contraceptive foam) up until the study completion, which will take a total of 30 days. Participation in a research study or use of an investigational drug in the last two months.
* An employee or student under supervision of any of the investigators of this study.
* Individuals who cannot state a good understanding of this study including risks and requirements; are unable to follow the rules of this study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Bioequivalence using pharmacokinetic endpoint of peak blood concentration (Cmax). | 24 hours
  Ten blood samples (10 mL) will be obtained at zero time (baseline) and at 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours after oral administration of 5 mg capsule of tacrolimus. Each healthy volunteer will be given a single oral dose of tacrolimus, 5 mg, on four separate occasions with at least a 2 week washout between study days. The peak exposure will be assessed by measuring the peak blood concentration (Cmax) obtained directly from the data. The treatment arms (aged Prograf®, fresh generic, aged generic) will be compared to fresh Prograf®. If the 90% confidence interval for the ratio of the measures in the treatment arms to the fresh Prograf is within the limits of 0.8 to 1.25 for the Cmax, the treatment measures will be judged bioequivalent.
Bioequivalence using pharmacokinetic endpoints of the area under the blood concentration vs time curve (AUC). | 24 hours
  Ten blood samples (10 mL) will be obtained at zero time (baseline) and at 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours after oral administration of 5 mg capsule of tacrolimus. Each healthy volunteer will be given a single oral dose of tacrolimus, 5 mg, on four separate occasions with at least a 2 week washout between study days. The AUC will be computed using the linear trapezoidal rule. The total exposure will be assessed by comparing the AUC from zero to 24 hours and the AUC from zero to infinity. The treatment arms (aged Prograf®, fresh generic, aged generic) will be compared to fresh Prograf®. If the 90% confidence interval for the ratio of the measures in the treatment arms to the fresh Prograf is within the limits of 0.8 to 1.25 for the AUC, the treatment measures will be judged bioequivalent.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond E Galinsky, PharmD, Principal Investigator — Indiana University; Brian Decker, MD, PharmD, Principal Investigator — Indiana University; Lynne S Taylor, PhD, Principal Investigator — Purdue University
Locations (1):
- Indiana CTSI Clinical Research Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fahr A, Liu X. Drug delivery strategies for poorly water-soluble drugs. Expert Opin Drug Deliv. 2007 Jul;4(4):403-16. doi: 10.1517/17425247.4.4.403. PMID 17683253
- [Result] Hancock BC, Parks M. What is the true solubility advantage for amorphous pharmaceuticals? Pharm Res. 2000 Apr;17(4):397-404. doi: 10.1023/a:1007516718048. PMID 10870982
- [Result] Kwong AD, Kauffman RS, Hurter P, Mueller P. Discovery and development of telaprevir: an NS3-4A protease inhibitor for treating genotype 1 chronic hepatitis C virus. Nat Biotechnol. 2011 Nov 8;29(11):993-1003. doi: 10.1038/nbt.2020. PMID 22068541
- [Result] Rumondor AC, Stanford LA, Taylor LS. Effects of polymer type and storage relative humidity on the kinetics of felodipine crystallization from amorphous solid dispersions. Pharm Res. 2009 Dec;26(12):2599-606. doi: 10.1007/s11095-009-9974-3. Epub 2009 Oct 6. PMID 19806435
- [Result] Baird JA, Taylor LS. Evaluation of amorphous solid dispersion properties using thermal analysis techniques. Adv Drug Deliv Rev. 2012 Apr;64(5):396-421. doi: 10.1016/j.addr.2011.07.009. Epub 2011 Aug 4. PMID 21843564
- [Result] Zucman D, Camara S, Gravisse J, Dimi S, Vasse M, Goudjo A, Choquet M, Peytavin G. Generic antiretroviral drugs in developing countries: friends or foes? AIDS. 2014 Feb 20;28(4):607-9. doi: 10.1097/QAD.0000000000000170. PMID 24378755
- [Result] Petan JA, Undre N, First MR, Saito K, Ohara T, Iwabe O, Mimura H, Suzuki M, Kitamura S. Physiochemical properties of generic formulations of tacrolimus in Mexico. Transplant Proc. 2008 Jun;40(5):1439-42. doi: 10.1016/j.transproceed.2008.03.091. PMID 18589125
- [Result] Momper JD, Ridenour TA, Schonder KS, Shapiro R, Humar A, Venkataramanan R. The impact of conversion from prograf to generic tacrolimus in liver and kidney transplant recipients with stable graft function. Am J Transplant. 2011 Sep;11(9):1861-7. doi: 10.1111/j.1600-6143.2011.03615.x. Epub 2011 Jun 30. PMID 21714845
- [Result] Pasqualotto AC, Denning DW. Generic substitution of itraconazole resulting in sub-therapeutic levels and resistance. Int J Antimicrob Agents. 2007 Jul;30(1):93-4. doi: 10.1016/j.ijantimicag.2006.11.027. Epub 2007 Apr 6. No abstract available. PMID 17412566
- [Result] Calahan JL, Zanon RL, Alvarez-Nunez F, Munson EJ. Isothermal microcalorimetry to investigate the phase separation for amorphous solid dispersions of AMG 517 with HPMC-AS. Mol Pharm. 2013 May 6;10(5):1949-57. doi: 10.1021/mp300714g. Epub 2013 Apr 24. PMID 23574401
- [Result] Pham TN, Watson SA, Edwards AJ, Chavda M, Clawson JS, Strohmeier M, Vogt FG. Analysis of amorphous solid dispersions using 2D solid-state NMR and (1)H T(1) relaxation measurements. Mol Pharm. 2010 Oct 4;7(5):1667-91. doi: 10.1021/mp100205g. Epub 2010 Aug 3. PMID 20681586